CLINICAL TRIAL: NCT07349693
Title: A Randomized Trial to Assess the Efficacy and Safety of Cerebraca Wafer Plus Temozolomide Versus Temozolomide Alone in Recurrent Glioblastoma
Brief Title: Comparison of Cerebraca Wafer Plus Temozolomide Versus Temozolomide Alone in Recurrent Glioblastoma
Acronym: Cerebraca-02/3
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Everfront Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFBPOLZ-1
Record Dates: First submitted 2026-01-15; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Glioblastoma, IDH-Wildtype
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Cerebraca Wafer) (Experimental): Patients will receive surgical tumor resection, implantation of 6 Cerebraca Wafer (75 mg each, total dose of 450 mg (Z)-BP) at the time of surgery, followed by SOC TMZ therapy.
  Interventions: Drug: Cerebraca wafer; Drug: Temozolomide (for relapsed malignant glioma)
- Comparative Group (Standard-of-Care) (Active Comparator): Patients will receive surgical tumor resection, followed by SOC TMZ therapy.
  Interventions: Drug: Temozolomide (for relapsed malignant glioma)

INTERVENTIONS:
Drug: Cerebraca wafer — Cerebraca Wafer, (75 mg (Z)-n-butylidenephthalide, (Z)-BP, Implant)
  Arms: Treatment Group (Cerebraca Wafer)
Drug: Temozolomide (for relapsed malignant glioma) — TMZ as the standard-of-care (SOC) treatment for recurrent glioblastoma.

SUMMARY:
This study is designed as a multi-center, randomized, open-label trial to evaluate the efficacy of Cerebraca Wafer in patients with recurrent glioblastoma. Cerebraca Wafer is intended for use in recurrent glioblastoma as an adjunct to surgery (followed by standard-of-care temozolomide), demonstrating potential to improve outcomes in this serious and life-threatening condition

ELIGIBILITY:
Inclusion Criteria, subjects must meet all following criteria for study enrollment:

1. Subject must be aged ≥ 18, regardless of gender
2. Subject must have histologically confirmed glioblastoma with:

   1. Completed first-line therapy including surgery plus temozolomide and radiation (concurrent temozolomide/radiation)
   2. Current presentation being first or second recurrence only
3. Subject must have measurable disease preoperatively with at least one contrast-enhancing MRI-identified lesion measuring ≥ 1 cm in two perpendicular dimensions per RANO 2.0 criteria
4. Subject must be deemed eligible for gross total resection of contrast-enhancing MRI-identified lesion by neurosurgeon's pre-operative assessment, according to RANO II
5. Subject must have Karnofsky Performance Status (KPS) ≥ 70
6. Subject must have recovered from prior therapy toxicities with adequate organ function:

   1. Hemoglobin ≥ 8 g/dL
   2. Platelets ≥ 100,000/mm3
   3. White blood cell count (WBC) ≥ 3,000 cells/mm3
   4. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
   5. Absolute lymphocyte count (ALC) ≥ 1,000 cells/mm3
   6. Coagulation tests (prothrombin time [PT], activated partial thromboplastin time [APTT], International Normalized Ratio [INR]) ≤ 1.5 × ULN
   7. Total bilirubin (TBIL) < 3 × ULN
   8. Alkaline phosphatase (ALP) ≤ 3 × ULN and/or Gamma glutamyltransferase (GGT) ≤ 1.5 × ULN
   9. Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and/or Alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 3 x ULN
   10. eGFR ≥ 30 mL/min (MDRD formula)
   11. QTc interval: msec ≤ 450 (males) or 470 (females) (Fridericia's formula: QTc=QT/RR(1/3); RR=RR interval)

Exclusion Criteria, subjects with any of the following will be excluded:

1. Histological confirmation of oligodendroglioma or mixed glioma
2. Presence of IDH or H3K27M mutation, or 1p19q co-deletion
3. MRI-identified lesion meeting any criteria:

   1. Multi-focal (defined as 2 non-contiguous contrast enhancement areas > 1 cm in 2 planes on fluid-attenuated inversion recovery, FLAIR or T2-weighted sequences)
   2. Presence of diffuse subependymal or leptomeningeal dissemination
   3. Contrast-enhancing lesion > 6 cm in any dimension
4. Tumor location unsuitable for surgical resection and Cerebraca Wafer implantation in the brain areas where surgical intervention would cause significant neurological deficits
5. Prior bevacizumab treatment with uncontrollable tumor progression
6. History of other malignancy within past 5 years
7. Immunocompromised status or autoimmune conditions requiring systemic immunosuppressive therapy, with the following exceptions:

   1. Patients with autoimmune conditions may be eligible after individual assessment of the condition, its severity, and potential interaction with the Cerebraca Wafer.
   2. Patients with HIV infection are eligible if they:

   i. Have CD4+ T-cell counts ≥350 cells/μL ii. Are on stable anti-retroviral therapy iii. Have HIV viral load below the limit of quantification c. Patients with HBV infection are eligible if they: i. Are on appropriate suppressive anti-viral therapy prior to study enrollment ii. Have no evidence of hepatic decompensation d. Patients with history of HCV infection are eligible if they: i. Have completed curative anti-viral treatment with HCV viral load below the limit of quantification
8. Active, uncontrolled infection or medical condition that could compromise safety and efficacy assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Median overall survival (OS) | 24 months
  Median overall survival (OS) in recurrent glioblastoma patients (event-based)

SECONDARY OUTCOMES:
Tolerability and Safety Profile | 24 months
  Number of participants with treatment-related adverse events and serious adverse events as assessed by CTCAE v5.0"
Survival rate | 6, 9, 12, 18, and 24 months
  To evaluate survival rate post resection.
Median progression-free survival (PFS) | 24 months
  To determine the median progression-free survival (PFS) in recurrent glioblastoma patients.
PFS rate | 6, 9, and 12 months
  To evaluate PFS rate at 6, 9, and 12 months post resection

CONTACTS AND LOCATIONS:
Locations (1):
- Legorreta Cancer Center Warren Alpert Medical School of Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes